CLINICAL TRIAL: NCT03267095
Title: The Use Of Music Therapy In Autism Spectrum Disorder
Brief Title: Use Music Therapy In Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mylove Amira, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTH ASD
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): .Patient in stduy Arm will receive music therapy sessions
  Interventions: Behavioral: music therapy sessions .
- Control (No Intervention): Patient in control Arm will have cosuling for mother and follow up

INTERVENTIONS:
Behavioral: music therapy sessions . — In this intervention songs compose by the therapist will be use for the study. The songs included the target word .The target words will be selecte from functional vocabularies that typically developing 3years old children can use effectively in everyday interactions.The general criteria for vocabulary words included: names of familiar objects and persons, functional action words such as words for social control , and emotional words . Inherent musical structures structures and organized musical patterns in the songs will be provide .The patients will reflect on the music therapy activity as singing the song together.
  Arms: Study

SUMMARY:
Music therapy is an established form of creative art therapy. By using music as a specific medium of communication, expression and adapting it to the individual resources and abilities of the patient, music therapy can be beneficial in activating and supporting mental and psycho-physical recover .

DETAILED DESCRIPTION:
Students with developmental disabilities often have challenges in the areas of communication and social/emotional learning, which can lead to social isolation, problematic behaviors, and deficits in academic learning.These students have been found to respond well to the incorporation of music in intervention programs, in terms of both gains in communication skills and stronger social functioning . they respond more favorably and appropriately to music than other sensory stimuli

ELIGIBILITY:
Inclusion Criteria:

* 1.Age :3_7 2.Gender : both sex will be included in the study 3.IQ ≥75 4.children who will dignosed by an expert phoniatricist as having ASD

Exclusion Criteria:

* 1.Age >3 <7 2.IQ <75 . 3. children having other cause of DELAYED LANGUAGE DEVELOPMENT

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
The Arabic Language test | Baseline,Change from Baseline at the end of 12 Months Music Therapy .
  The Arabic Language test:
  language score is the sum of the total scores of: Test of semantics Test of expressive morphology Test of syntax Test of pragmatics

REFERENCES:
- [Background] Gold C, Voracek M, Wigram T. Effects of music therapy for children and adolescents with psychopathology: a meta-analysis. J Child Psychol Psychiatry. 2004 Sep;45(6):1054-63. doi: 10.1111/j.1469-7610.2004.t01-1-00298.x. PMID 15257662
- [Derived] Geretsegger M, Fusar-Poli L, Elefant C, Mossler KA, Vitale G, Gold C. Music therapy for autistic people. Cochrane Database Syst Rev. 2022 May 9;5(5):CD004381. doi: 10.1002/14651858.CD004381.pub4. PMID 35532041